CLINICAL TRIAL: NCT06729268
Title: Possibility of Applying Fluid Responsiveness Tests in Critically Ill Patients During Admission to the Intensive Care Unit - a Prospective Observational Study.
Brief Title: Fluid Responsiveness Tests in Critically Ill Patients During Admission to the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Ryszard Gawda, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Other Study IDs: PossFluRespTests
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Shock Circulatory; Heart Failure; Hypovolemia
MeSH Terms: conditions — Shock; Heart Failure; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated in the intensive care unit: Patients treated in the intensive care unit during the first six hours after admission.

SUMMARY:
The goal of this observational study is to investigate the prevalence of conditions allowing the performance fluid responsiveness tests in critically ill patients during admission to the intensive care unit.

DETAILED DESCRIPTION:
Patients admitted to the intensive care unit are very often hemodynamically unstable. In these cases fluid responsiveness tests should be performed to assess whether the patient would benefit from the fluid administration.

However, fluid responsiveness tests have many limitations including lack of spontaneous breathing, necessity of invasive mechanical ventilation with tidal volume of > 8 mL/kg ideal body weight, regular hearth rhythm, and lack of abdominal hypertension.

In the study, the investigators evaluated the prevalence of conditions enabling the performance fluid responsiveness tests in patients admitted to the intensive care unit. An assessment was performed within the six hours after admission to the intensive care unit. Evaluation was based on transthoracic echocardiography, clinical examination of the patients, and data derived from anamnesis.

The following fluid responsiveness tests were included into assessment: passive leg raising test, end-expiratory occlusion test, pulse pressure variation, stroke volume variation, velocity time integral variation in left ventricle output track, tidal volume challenge, inferior vena cava diameter variation, and superior vena cava diameter variation.

The aim of the study was to assess how many patients have the conditions allowing performance fluid responsiveness tests during admission to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients admitted to the intensive care unit

Exclusion Criteria:

1. Age under 18
2. The researcher unavailable in the intensive care unit
3. Patient assessment cannot be completed within the first six hours after admission to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of conditions allowing the performance fluid responsiveness tests during admission to the intensive care unit. | Six hours after admission to the intensive care unit
  The primary aim of the study is to assess the prevalence of conditions allowing the performance fluid responsiveness tests during admission to the intensive care unit.

SECONDARY OUTCOMES:
To assess which fluid responsiveness test based on heart-lung interactions can be applied most often during admission to the intensive care unit | Six hours after admission to the intensive care unit
  The secondary aim of the study is to assess which fluid responsiveness test based on heart-lung interaction can be applied most often during admission to the intensive care unit
To assess the percentage of patients in shock whom fluid responsiveness tests can be performed during admission to the intensive care unit | Six hours from the admission to the intensive care unit.
  Secondary aim include an assessment the percentage of patients in shock whom fluid responsiveness tests can be performed during admission to the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No